CLINICAL TRIAL: NCT00771667
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Ustekinumab Therapy in Subjects With Moderately to Severely Active Crohn's Disease Previously Treated With TNF Antagonist Therapy
Brief Title: A Study of Safety and Effectiveness of Ustekinumab in Patients With Moderate to Severe Active Crohn's Disease Who Have Been Previously Treated With Anti-TNF Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Director, Clinical Research, Janssen R&D US
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015238; C0743T26 (Other: Centocor)
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Interleukin-12; Inflammation; Research study; Ustekinumab; CNTO1275; Interleukin-23
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Placebo (IP) (Placebo Comparator)
  Interventions: Drug: Placebo (IP)
- Ustekinumab 1mg/kg (IP) (Experimental)
  Interventions: Drug: Ustekinumab 1mg/kg (IP)
- Ustekinumab 3 mg/kg (IP) (Experimental)
  Interventions: Drug: Ustekinumab 3 mg/kg (IP)
- Ustekinumab 6 mg/kg (IP) (Experimental)
  Interventions: Drug: Ustekinumab 6 mg/kg (IP)
- Placebo IV - Responder - Placebo SC (MP) (Placebo Comparator)
  Interventions: Drug: Placebo IV - Responder - Placebo SC (MP)
- Placebo IV - Nonresponder - Ustekinumab 270/90 mg SC (Placebo Comparator)
  Interventions: Drug: Placebo IV - Nonresponder - Ustekinumab 270/90 mg SC (MP)
- Ustekinumab IV - Responder - Placebo SC (MP) (Placebo Comparator)
  Interventions: Drug: Ustekinumab IV - Responder - Placebo SC (MP)
- Ustekinumab IV - Responder - Ustekinumab 90mg SC (MP) (Experimental)
  Interventions: Drug: Ustekinumab IV - Responder - Ustekinumab 90mg SC (MP)
- Ustekinumab IV - Nonresponder - Placebo SC (MP) (Placebo Comparator)
  Interventions: Drug: Ustekinumab IV - Nonresponder - Placebo SC (MP)
- Ustekinumab IV - Nonresponder - Ustekinumab 90mg SC (MP) (Experimental)
  Interventions: Drug: Ustekinumab IV - Nonresponder - Ustekinumab 90mg SC (MP)

INTERVENTIONS:
Drug: Placebo (IP) — Induction phase (Week 0-8) (IP) - Placebo IV group
  Arms: Placebo (IP)
Drug: Ustekinumab 1mg/kg (IP) — Induction phase (Week 0-8) (IP) - Ustekinumab 1 mg/kg IV group
  Arms: Ustekinumab 1mg/kg (IP)
Drug: Ustekinumab 3 mg/kg (IP) — Induction phase (Week 0-8) (IP) - Ustekinumab 3mg/kg IV group
  Arms: Ustekinumab 3 mg/kg (IP)
Drug: Ustekinumab 6 mg/kg (IP) — Induction phase (Week 0-8) (IP) - Ustekinumab 6mg/kg IV group
  Arms: Ustekinumab 6 mg/kg (IP)
Drug: Placebo IV - Responder - Placebo SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Placebo IV at Week 0 - Responder at week 6 - Receiving Placebo SC at Week 8 and Week 16
  Arms: Placebo IV - Responder - Placebo SC (MP)
Drug: Placebo IV - Nonresponder - Ustekinumab 270/90 mg SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Placebo IV at Week 0 - Nonresponder at week 6 - Receiving Ustekinumab 270 mg SC at Week 8 and 90 mg at Week 16
  Arms: Placebo IV - Nonresponder - Ustekinumab 270/90 mg SC
Drug: Ustekinumab IV - Responder - Placebo SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 - Responder at week 6 - Receiving Placebo SC at Week 8 and Week 16
  Arms: Ustekinumab IV - Responder - Placebo SC (MP)
Drug: Ustekinumab IV - Responder - Ustekinumab 90mg SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 - Responder at week 6 - Receiving Ustekinumab 90 mg SC at Week 8 and Week 16
  Arms: Ustekinumab IV - Responder - Ustekinumab 90mg SC (MP)
Drug: Ustekinumab IV - Nonresponder - Placebo SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 - Nonresponder at week 6 - Receiving Placebo SC at Week 8 and Week 16
  Arms: Ustekinumab IV - Nonresponder - Placebo SC (MP)
Drug: Ustekinumab IV - Nonresponder - Ustekinumab 90mg SC (MP) — Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 - Nonresponder at week 6 - Receiving Ustekinumab 90 mg SC at Week 8 and Week 16
  Arms: Ustekinumab IV - Nonresponder - Ustekinumab 90mg SC (MP)

SUMMARY:
A medical research study in adult patients who have moderate to severe Crohn's disease designed to determine whether or not treatment with an experimental drug called ustekinumab (or CNTO1275) is safe or not and to determine if the treatment will reduce the symptoms of Crohn's disease.

DETAILED DESCRIPTION:
In Crohn's disease there is inflammation (changes in body tissue which normally happen during injury or infection) and or ulceration (open sores) in the intestines.This occurs because the immune system (the part of the body that fights off infection) has an abnormal and overactive response against the intestine and bowel tissues of the body. Crohn's disease is usually treated with medications that either directly decrease inflammation or decrease the general activity of the immune system to improve the diarrhea, abdominal pain, and other symptoms of Crohn's Disease. Ustekinumab antibodies (natural substances made by your immune system to stick to and help remove foreign materials in your body that cause diseases) have been created to stick to and block the activity of two of the immune substances thought to cause abnormal inflammation of Crohn's disease. Patients who are eligible and who have received Remicade, Humira, or Cimzia and failed or been intolerant to one of these drugs will be randomized to either active drug (ustekinumab) or placebo. All patients will be randomized (like flipping a coin) at week 0 to be in one of 4 groups. At week 0 the study drug will be given by IV administration and at weeks 8 and 16 by subcutaneous injection. There will be 11 study visits in total and the study will continue until week 36. Blood and stool samples will be collected and studied, questionnaires to check on how you are doing in terms of your disease will be completed, an Electrocardiogram (EKG) obtained, safety evaluations conducted and diary cards distributed to be completed during the entire study. One of 4 groups: Grp 1-placebo, Grp 2-active drug 1mg/kg IV, Grp 3-active drug 3mg/kg IV, Grp 4-active drug 6mg/kg IV. Based on the clinical response status at Week 6, patients from Grps 2, 3 and 4 will be re-randomized at week 8 to receive either placebo or 90 mg SC at both weeks 8 and 16 and patients from Grp 1 will receive placebo at Week 8 and Week 16 or a 270 mg SC injection at Week 8 and 90 mg SC at Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Must have Crohn's disease or fistulizing Crohn's disease of at least 3 months duration
* Must have received Remicade, adalimumab or Cimzia at a dose approved for the treatment of Crohn's disease
* Must have failed or been intolerant to Remicade, Humira or Cimzia for treatment of Crohn's disease
* Must be 18 years of age or older
* Must have active Crohn's disease according to the Crohn's Disease Activity Index (CDAI > =220 and < =450).

Exclusion Criteria:

* Patients who have had any kind of bowel resection, diversions or placement of a stoma within 6 months
* Are pregnant, nursing or planning pregnancy (both men and women) while enrolled in the study or within 1 year after receiving study agent
* Patients who have received Remicade, Humira or Cimzia < =8 weeks before the first administration of study drug
* Patients with certain complications of Crohn's disease that would make it hard to assess response to study drug
* Patients with a history of or ongoing chronic or recurrent infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (174):
- United States (88):
  - Mobile, Alabama
  - Scottsdale, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Roseville, California
  - San Carlos, California
  - San Francisco, California
  - Englewood, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Hamden, Connecticut
  - Gainesville, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Port Charlotte, Florida
  - Port Orange, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Newnan, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Clive, Iowa
  - Pratt, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Detroit, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Ocean Springs, Mississippi
  - Mexico, Missouri
  - Lebanon, New Hampshire
  - Egg Harbor, New Jersey
  - Great Neck, New York
  - New York, New York
  - Poughkeepsie, New York
  - Setauket, New York
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Kinston, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Beavercreek, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Lewisville, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Bellevue, Washington
  - Lakewood, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
- Australia (14):
  - Adelaide
  - Bankstown
  - Bedford Park
  - Box Hill
  - Concord
  - East Melbourne
  - Fitzroy
  - Frankston
  - Fremantle
  - Garran
  - Herston
  - Parkville
  - Prahran
  - South Brisbane
- Austria (4):
  - Innsbruck
  - Linz
  - Salzburg
  - Vienna
- Belgium (7):
  - Bonheiden
  - Brussels
  - Edegem
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- France (8):
  - Amiens Cedex 1 80
  - Grenoble
  - Lille
  - Nice
  - Paris
  - Pessac
  - Rouen
  - Toulouse Cedex 9 N/A
- Germany (11):
  - Berlin
  - Hamburg
  - Hanover
  - Kiel
  - Leipzig
  - Lÿneburg
  - Markkleeberg
  - Minden
  - München
  - Münster
  - Regensburg
- Israel (7):
  - Afula
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Tel Aviv
- Netherlands (5):
  - Amersfoort
  - Amsterdam
  - Leiden
  - Maastricht
  - Rotterdam
- New Zealand (2):
  - Auckland
  - Christchurch
- Spain (8):
  - Barcelona
  - Córdoba
  - León
  - Madrid
  - Oviedo
  - Palma
  - Sabadell
  - Zaragoza
- United Kingdom (10):
  - Bristol
  - Cambridge
  - Coventry
  - Edinburgh
  - Harrow
  - London
  - Manchester
  - Newcastle upon Tyne
  - Norwich
  - Nottinghamshirecc

REFERENCES:
- [Derived] Adedokun OJ, Xu Z, Gasink C, Kowalski K, Sandborn WJ, Feagan B. Population Pharmacokinetics and Exposure-Response Analyses of Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease. Clin Ther. 2022 Oct;44(10):1336-1355. doi: 10.1016/j.clinthera.2022.08.010. Epub 2022 Sep 21. PMID 36150926
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Di Narzo AF, Telesco SE, Brodmerkel C, Argmann C, Peters LA, Li K, Kidd B, Dudley J, Cho J, Schadt EE, Kasarskis A, Dobrin R, Hao K. High-Throughput Characterization of Blood Serum Proteomics of IBD Patients with Respect to Aging and Genetic Factors. PLoS Genet. 2017 Jan 27;13(1):e1006565. doi: 10.1371/journal.pgen.1006565. eCollection 2017 Jan. PMID 28129359
- [Derived] Sandborn WJ, Gasink C, Gao LL, Blank MA, Johanns J, Guzzo C, Sands BE, Hanauer SB, Targan S, Rutgeerts P, Ghosh S, de Villiers WJ, Panaccione R, Greenberg G, Schreiber S, Lichtiger S, Feagan BG; CERTIFI Study Group. Ustekinumab induction and maintenance therapy in refractory Crohn's disease. N Engl J Med. 2012 Oct 18;367(16):1519-28. doi: 10.1056/NEJMoa1203572. PMID 23075178

RESULTS

PARTICIPANT FLOW:
Groups:
- Ustekinumab 1 mg/kg (IP): Induction phase (Week 0-8) (IP) - Ustekinumab 1mg/kg IV group
- Placebo IV -> Responder -> Placebo SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Placebo IV at Week 0 -> Responder at week 6 -> Receiving Placebo SC at Week 8 and Week 16
- Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Placebo IV at Week 0 -> Nonresponder at week 6 -> Receiving Ustekinumab 270 mg SC at Week 8 and 90 mg at Week 16
- Ustekinumab IV -> Responder -> Placebo SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 -> Responder at week 6 -> Receiving Placebo SC at Week 8 and Week 16
- Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 -> Responder at week 6 -> Receiving Ustekinumab 90 mg SC at Week 8 and Week 16
- Ustekinumab IV -> Nonresponder -> Placebo SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 -> Nonresponder at week 6 -> Receiving Placebo SC at Week 8 and Week 16
- Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP): Maintenance phase (Week 8-36) (MP) - Receiving Ustekinumab IV at Week 0 -> Nonresponder at week 6 -> Receiving Ustekinumab 90 mg SC at Week 8 and Week 16
Period: Induction Phase
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP) | Placebo IV -> Responder -> Placebo SC (MP) | Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP) | Ustekinumab IV -> Responder -> Placebo SC (MP) | Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP) | Ustekinumab IV -> Nonresponder -> Placebo SC (MP) | Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP)
Started | 132 | 131 | 132 | 131 | 0 ("0" in column indicates this reporting group is not relevant to Induction period.) | 0 ("0" in column indicates this reporting group is not relevant to Induction period.) | 0 ("0" in column indicates this reporting group is not relevant to Induction period.) | 0 ("0" in column indicates this reporting group is not relevant to Induction period.) | 0 ("0" in column indicates this reporting group is not relevant to Induction period.) | 0 ("0" in column indicates this reporting group is not relevant to Induction period.)
Completed | 113 | 121 | 120 | 123 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 19 | 10 | 12 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 6 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP) | Placebo IV -> Responder -> Placebo SC (MP) | Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP) | Ustekinumab IV -> Responder -> Placebo SC (MP) | Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP) | Ustekinumab IV -> Nonresponder -> Placebo SC (MP) | Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP)
Started | 0 ("0" in column indicates this reporting group is not relevant to Maintenance period.) | 0 ("0" in column indicates this reporting group is not relevant to Maintenance period.) | 0 ("0" in column indicates this reporting group is not relevant to Maintenance period.) | 0 ("0" in column indicates this reporting group is not relevant to Maintenance period.) | 28 | 85 | 73 | 72 | 110 | 109
Completed | 0 | 0 | 0 | 0 | 26 | 78 | 63 | 67 | 88 | 92
Not Completed | 0 | 0 | 0 | 0 | 2 | 7 | 10 | 5 | 22 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 1 | 8 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 11 | 7
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP) | Total
Number analyzed (Participants) | 132 | 131 | 132 | 131 | 526
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.05) | 38.8 (11.95) | 38.2 (12.63) | 39.4 (13.21) | 39 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 83 | 75 | 83 | 309
  Male | 64 | 48 | 57 | 48 | 217

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Week 6
Description: As measured by the Crohn's Disease Activity Index (CDAI). CDAI scores range from 0 points (minimal disease activity) to over 600 points (severe disease activity). Clinical response was defined as a reduction from baseline of ≥ 100 points. Participants with a baseline CDAI of ≥ 220 to ≤ 248 were considered to be in clinical response if a CDAI score of < 150 was attained.
Time Frame: Baseline to Week 6
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP)
Number analyzed (Participants) | 132 | 131 | 132 | 131
Participants | 31 | 48 | 45 | 52
Statistical Analysis 1: Comparison: Placebo (IP) vs Ustekinumab 6 mg/kg (IP); Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — A fixed sequence testing procedure was employed to control the type I error rate at 0.05 level for the primary endpoint, beginning with the highest dose; The CMH test is controlling for anti-TNF status
Statistical Analysis 2: Comparison: Placebo (IP) vs Ustekinumab 3 mg/kg (IP); Test type: Superiority or Other; p = 0.057, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The CMH test is controlling for anti-TNF status
Statistical Analysis 3: Comparison: Placebo (IP) vs Ustekinumab 1 mg/kg (IP); Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The CMH test is controlling for anti-TNF status

2. Secondary Outcome: Number of Participants With Clinical Remission at Week 6
Description: As measured by a CDAI score of < 150 points.
Time Frame: Baseline to Week 6
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP)
Number analyzed (Participants) | 132 | 131 | 132 | 131
Participants | 14 | 21 | 21 | 16
Statistical Analysis 1: Comparison: Placebo (IP) vs Ustekinumab 6 mg/kg (IP); Test type: Superiority or Other; p = 0.682, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 2: Comparison: Placebo (IP) vs Ustekinumab 3 mg/kg (IP); Test type: Superiority or Other; p = 0.206, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 3: Comparison: Placebo (IP) vs Ustekinumab 1 mg/kg (IP); Test type: Superiority or Other; p = 0.196, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status

3. Secondary Outcome: Number of Participants With Clinical Response at Week 4
Description: As measured by the CDAI. Clinical response was defined as a reduction from baseline of ≥ 100 points. Participants with a baseline CDAI of ≥ 220 to ≤ 248 were considered to be in clinical response if a CDAI score of < 150 was attained.
Time Frame: Baseline to Week 4
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP)
Number analyzed (Participants) | 132 | 131 | 132 | 131
Participants | 22 | 36 | 49 | 40
Statistical Analysis 1: Comparison: Placebo (IP) vs Ustekinumab 6 mg/kg (IP); Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 2: Comparison: Placebo (IP) vs Ustekinumab 3 mg/kg (IP); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 3: Comparison: Placebo (IP) vs Ustekinumab 1 mg/kg (IP); Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status

4. Secondary Outcome: Number of Participants With Clinical Response at Week 8
Description: as for outcome 3
Time Frame: Baseline to Week 8
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP)
Number analyzed (Participants) | 132 | 131 | 132 | 131
Participants | 23 | 42 | 42 | 57
Statistical Analysis 1: Comparison: Placebo (IP) vs Ustekinumab 6 mg/kg (IP); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 2: Comparison: Placebo (IP) vs Ustekinumab 3 mg/kg (IP); Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 3: Comparison: Placebo (IP) vs Ustekinumab 1 mg/kg (IP); Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status

5. Secondary Outcome: Number of Participants With Clinical Remission at Week 8
Description: As measured by a CDAI score of < 150 points.
Time Frame: Baseline to Week 8
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP)
Number analyzed (Participants) | 132 | 131 | 132 | 131
Participants | 14 | 23 | 24 | 24
Statistical Analysis 1: Comparison: Placebo (IP) vs Ustekinumab 6 mg/kg (IP); Test type: Superiority or Other; p = 0.074, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 2: Comparison: Placebo (IP) vs Ustekinumab 3 mg/kg (IP); Test type: Superiority or Other; p = 0.081, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status
Statistical Analysis 3: Comparison: Placebo (IP) vs Ustekinumab 1 mg/kg (IP); Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel; The CMH test is controlling for anti-TNF status

6. Secondary Outcome: Number of Participants With Clinical Remission at Week 22 (Among Responders From Week 6)
Description: As measured by a CDAI score of < 150 points.
Time Frame: Baseline to Week 22
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Groups:
- Placebo SC; Ustekinumab 90 mg SC: As a single subcutaneous dose at Weeks 8 and 16
Arm/Group | Placebo SC | Ustekinumab 90 mg SC
Number analyzed (Participants) | 73 | 72
Participants | 20 | 30
Statistical Analysis 1: Comparison: Placebo SC vs Ustekinumab 90 mg SC; Test type: Superiority or Other; p = 0.029, Cochran-Mantel-Haenszel — Testing for Week-22 clinical remission was performed if the comparison of 6-mg/kg ustekinumab with placebo was positive for the primary endpoint; The CMH test chi-square test, stratified by IV induction dose and clinical remission status at Week 6

7. Secondary Outcome: Number of Participants With Clinical Response at Week 22 (Among Responders From Week 6)
Description: as for outcome 3
Time Frame: Baseline to Week 22
Population: All participants who were randomized, regardless of whether they received study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo SC | Ustekinumab 90 mg SC
Number analyzed (Participants) | 73 | 72
Participants | 31 | 50
Statistical Analysis 1: Comparison: Placebo SC vs Ustekinumab 90 mg SC; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The CMH test is controlling for induction dose and clinical remission status at Week 6

ADVERSE EVENTS:
Arm/Group | Placebo (IP) | Ustekinumab 1 mg/kg (IP) | Ustekinumab 3 mg/kg (IP) | Ustekinumab 6 mg/kg (IP) | Placebo IV -> Responder -> Placebo SC (MP) | Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP) | Ustekinumab IV -> Responder -> Placebo SC (MP) | Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP) | Ustekinumab IV -> Nonresponder -> Placebo SC (MP) | Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP)
Serious Adverse Events (participants affected / at risk) | 11/132 | 6/130 | 8/133 | 9/131 | 8/28 | 16/85 | 12/73 | 9/72 | 21/110 | 22/109
Other Adverse Events (participants affected / at risk) | 53/132 | 51/130 | 50/133 | 47/131 | 18/28 | 47/85 | 39/73 | 39/72 | 64/110 | 52/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (IP) (N=132) | Ustekinumab 1 mg/kg (IP) (N=130) | Ustekinumab 3 mg/kg (IP) (N=133) | Ustekinumab 6 mg/kg (IP) (N=131) | Placebo IV -> Responder -> Placebo SC (MP) (N=28) | Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP) (N=85) | Ustekinumab IV -> Responder -> Placebo SC (MP) (N=73) | Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP) (N=72) | Ustekinumab IV -> Nonresponder -> Placebo SC (MP) (N=110) | Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP) (N=109)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 5 | 2 | 4 | 2 | 3 | 8 | 7 | 4 | 8 | 10
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serum sickness-like reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anal abscess (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (IP) (N=132) | Ustekinumab 1 mg/kg (IP) (N=130) | Ustekinumab 3 mg/kg (IP) (N=133) | Ustekinumab 6 mg/kg (IP) (N=131) | Placebo IV -> Responder -> Placebo SC (MP) (N=28) | Placebo IV -> Nonresponder -> Ustekinumab 270/90 mg SC (MP) (N=85) | Ustekinumab IV -> Responder -> Placebo SC (MP) (N=73) | Ustekinumab IV -> Responder -> Ustekinumab 90mg SC (MP) (N=72) | Ustekinumab IV -> Nonresponder -> Placebo SC (MP) (N=110) | Ustekinumab IV -> Nonresponder -> Ustekinumab 90mg SC (MP) (N=109)
Abdominal pain (Gastrointestinal disorders) | 9 | 5 | 8 | 7 | 1 | 4 | 8 | 3 | 10 | 7
Crohn's disease (Gastrointestinal disorders) | 8 | 5 | 3 | 3 | 10 | 9 | 16 | 7 | 19 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 1 | 0 | 4 | 2 | 5 | 2
Nausea (Gastrointestinal disorders) | 11 | 9 | 1 | 8 | 3 | 8 | 5 | 7 | 8 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 3 | 0 | 2 | 4 | 6 | 6 | 5
Fatigue (General disorders) | 0 | 3 | 4 | 1 | 0 | 2 | 5 | 2 | 4 | 1
Pyrexia (General disorders) | 3 | 5 | 4 | 3 | 1 | 8 | 2 | 1 | 9 | 6
Nasopharyngitis (Infections and infestations) | 6 | 7 | 7 | 8 | 1 | 12 | 6 | 5 | 0 | 6
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 2 | 1 | 1 | 3 | 4 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 4 | 5 | 2 | 2 | 4 | 6 | 7 | 7
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 1 | 2 | 1 | 0 | 3 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 8 | 6 | 2 | 7 | 3 | 5 | 12 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4 | 4 | 2 | 2 | 3 | 3 | 6 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 6 | 3 | 0 | 1 | 4 | 2 | 3 | 1
Headache (Nervous system disorders) | 8 | 8 | 9 | 13 | 1 | 5 | 4 | 4 | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 4 | 3 | 4 | 2 | 4 | 1 | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 3 | 1 | 1 | 2 | 1 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days